CLINICAL TRIAL: NCT01169961
Title: Assessment of Iron Deposition in Major Organs of Hemodialysis Patients, Using T2*MRI and Novel Biomarkers of Free Iron Species
Brief Title: Assessment of Iron Deposition in Major Organs of Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Prof. E. Rachmilewitz, Head of Hematology in Wolfson Medical Center
Other Study IDs: 0003-10CTIL
Record Dates: First submitted 2010-07-23; First posted 2010-07-26 (Estimated); Last update posted 2010-07-26 (Estimated); Status verified 2010-07

CONDITIONS: Iron Overload
Keywords: IRON OVERLOAD IN HEMODIALYSIS PATIENTS
MeSH Terms: conditions — Iron Overload

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the present study is to evaluate in hemodialysis patients, who have elevated serum ferritin ( >2000ng/ml) and transferrin saturation (TSAT) >30%, iron deposition in the heart, pancreas, liver and spleen using the T2* MRI technique.

In addition, we will also measure the free iron forms in the plasma and LPI, LCI in red blood cells, platelets and PMN, in addition to serum hepcidin, TSAT, serum ferritin, CRP and oxidative stress parameters (ROS,GSH, and malonyldialdehyde (MDA).

DETAILED DESCRIPTION:
Despite the foregoing advances in the management of anemia associated with chronic kidney disease by the use of erythropoiesis stimulating agents and intravenous iron, assessment of iron status in these patients remains an unresolved issue.

It is estimated that following administration of erythropoietin together with intravenous iron, nearly 50% of all hemodialysis patients in the United states have a serum ferritin >500ng/ml (1). However, in many patients high serum ferritin levels (>2000ng/ml) have been documented. These levels are indicative of iron overload, also defined as hemosiderosis (2).

The risk of using IV iron in spite of serum ferritin levels of >2000ng/ml can result in accumulation of excess iron in tissues, such as the heart, liver, and pancreas similar to findings in patients with hemochromatosis (3) with possible deleterious effects. Accordingly, a recent study indicated a mathematically significant correlation between serum ferritin and liver iron stores using the indirect imaging known as SQUID (4).

Recently, T2*MRI (magnetic resonance imaging) became a non-invasive modality for evaluating tissue iron stores (5). Since high iron content shortens the T2* relaxation, decreased T2* values have been advocated as an early marker of iron deposition in target organs, related to the paramagnetic properties of hemosiderosis (5). This method is commonly used to evaluate and monitor iron deposition in major organs in thalassemia major and myelodysplastic syndrome (MDS) who are multitransfused.

In the former diseases, one of the consequences of iron overload is the presence of labile iron forms, which are redox active and therefore are associated with the propensity to catalyze the generation of reactive oxygen species (ROS) by the Haber Weiss reaction .Two forms of labile iron have been identified, one in the plasma (Labile plasma iron-LPI) and the other is found in the cells (labile cellular iron -LCI)(6,7 ).

In iron overload syndromes such as hemochromatosis, thalassemia or MDS these labile iron forms are increased, causing increased generation of oxidative stress with subsequent damage to membrane, cytoplasmatic and nuclear components.

An important master regulator of iron hemostasis is hepcidin, which is liver derived acute phase protein, and its synthesis is regulated by cytokines and iron status in the body (8).

It has been suggested that increased hepcidin levels may also contribute significantly to the severity of anemia of CKD.

ELIGIBILITY:
Inclusion Criteria:

* patients for study are > 50 years of age,
* on chronic hemodialysis for at least one year,
* with serum ferritin levels > 2000 ng/ml and TSAT > 30%.

Exclusion Criteria:

* malignancies,
* any active infection requiring systemic antibiotic therapy, and
* hospitalization within the two weeks before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hemodialysis patients, who have elevated serum ferritin ( >2000ng/ml) and transferrin saturation (TSAT) >30%
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
T2*MRI (magnetic resonance imaging) | one year
  This method is commonly used to evaluate and monitor iron deposition in major organs (iron overload) in hemodialysis patients with end stage renal failure

SECONDARY OUTCOMES:
Iron parameters (FERRITIN, TRANSFERREN SAT ,LPI HEPCIDIN,LCI,CRP,OXIDATIVE STRESS PARAMETERS(ROS,GSH,MDA) | ONE YEAR
  we will also measure the free iron forms in the plasma and LPI, LCI in red blood cells, platelets and PMN, in addition to serum hepcidin, TSAT, serum ferritin, CRP and oxidative stress parameters (ROS,GSH, and malonyldialdehyde (MDA).

CONTACTS AND LOCATIONS:
Overall Officials: GHOTI HOSSAM, Principal Investigator — HEMATOLOGY DEPARTMENT ON WOLFSSON MEDICAL CENTER
Locations (1):
- Wolfsson Medical Center, Holon, Israel, Israel